CLINICAL TRIAL: NCT01357538
Title: Efficacy and Safety of Posiformin 2 % Eye Ointment in the Treatment of Blepharitis - a Multi-centre, Randomised, Double-masked, Parallel-group, Phase IV Comparison
Brief Title: Efficacy and Safety of Posiformin 2 % Eye Ointment in the Treatment of Blepharitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ursapharm Arzneimittel GmbH (Industry)
Responsible Party: Prof. P. A. Bezdetko, Kharkov District Clincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: POFOBLE; S67-OPH-081; S67-OPH-081 (Other: RPS Germany)
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Blepharitis; Signs and Symptoms
Keywords: Bibrocathol; eye ointment; blepharitis; eye lid
MeSH Terms: conditions — Blepharitis; Signs and Symptoms | interventions — bibrocathol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Posiformin 2 % (Active Comparator): Eye ointment applied to the eye lid
  Interventions: Drug: Posiformin 2 %, bibrocathol
- Placebo (Placebo Comparator): corresponding vehicle, eye ointment applied to the eye lid
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Posiformin 2 %, bibrocathol — A strip of 5 mm eye ointment applied 3 times per day to the eye lid
  Arms: Posiformin 2 %
Drug: Placebo Comparator — corresponding vehicle, eye ointment applied to the eye lid
  Arms: Placebo

SUMMARY:
This is a multicentre, randomised, double-masked, parallel-group, phase IV comparison of Posiformin 2 % eye ointment (active substance: bibrocathol) in the treatment of blepharitis.

DETAILED DESCRIPTION:
Reduction of signs and symptoms of blepharitis

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* ambulatory male and female patients 18 years of age or older
* summarised score of signs and symptoms of blepharitis of 15 or more at baseline

Exclusion Criteria:

* different ocular conditions
* different system conditions
* several concomitant medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of Posiformin 2% in reduction of signs and symptoms of blepharitis | 14 days
  Changes from baseline in the sumscore which comprises lid edema, lid erythema, debris, pouting of Meibomian glands by slit lamp examination

SECONDARY OUTCOMES:
Changes in blepharitis signs and symptoms | 14 days
  Changes between baseline and end of treatment in lid edema, lid erythema, debris, pouting of meibomian glands, ocular discomfort, antiseptic effect

CONTACTS AND LOCATIONS:
Overall Officials: Pavel A Bezdetko, Prof., Principal Investigator — Kharkov District Clinical Hospital
Locations (1):
- Kharkov District Clinical Hospital, Kharkiv, Ukraine

REFERENCES:
- [Derived] Bezdetko PA, Sergienko N, Dyomin Y, Korol A, Nikitin N, Merzbacher M, Gross D, Kohnen R. Successful treatment of blepharitis with bibrocathol (Posiformin(R) 2 %). Graefes Arch Clin Exp Ophthalmol. 2012 Dec;250(12):1869-75. doi: 10.1007/s00417-012-2001-0. Epub 2012 Apr 25. PMID 22527308